CLINICAL TRIAL: NCT01477112
Title: Effect of the Supplementation With β-carotene to Type 2 Diabetic Patients and Healthy Controls on the Iron Status and Antioxidant Capacity of Plasma
Brief Title: Low Dose β-carotene Supplementation Diminishes Oxidative Stress in Type 2 Diabetics and Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Venezolano de Investigaciones Cientificas (Other)
Collaborators: Seguros Caracas Foundation (Unknown); National Fund for Science and Technology, Science Mission (Unknown)
Responsible Party: Principal Investigator, Maria Nieves Garcia-Casal, Director of Pathophysiology Laboratory, Instituto Venezolano de Investigaciones Cientificas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IVIC-HUMNUT-001
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus; Oxidative Stress; Iron Metabolism Disorders
Keywords: Type 2 diabetes; β-carotene; Oxidative balance; Oxidants; Antioxidants
MeSH Terms: conditions — Diabetes Mellitus; Iron Metabolism Disorders; Diabetes Mellitus, Type 2 | interventions — beta Carotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Supplemented Diabetics (DB) (Experimental): Diabetics supplemented with betacarotene for 45 days
  Interventions: Dietary Supplement: Betacarotene
- Unsupplemented Diabetics (DS) (Experimental): Diabetics without betacarotene supplementation
  Interventions: Dietary Supplement: Controls. No treatment
- Supplemented Controls (CB) (Active Comparator): Controls supplemented with betacarotene for 45 days
  Interventions: Dietary Supplement: Betacarotene
- Unsupplemented Controls (CS) (Active Comparator): Controls without betacarotene supplementation
  Interventions: Dietary Supplement: Controls. No treatment

INTERVENTIONS:
Dietary Supplement: Betacarotene — 6 mg betacarotene in caplets for 45 days (daily)and reevaluate parameters 30 days after finishing supplementation
  Other Names: β-carotene as a soft gel capsule (GNC, Pennsylvania-USA)
  Arms: Supplemented Controls (CB); Supplemented Diabetics (DB)
Dietary Supplement: Controls. No treatment — Evaluate at time 0, 45 days and 75 days, but without receiving betacarotene supplements
  Other Names: No supplements
  Arms: Unsupplemented Controls (CS); Unsupplemented Diabetics (DS)

SUMMARY:
Since diabetes has multiple etiologies and oxidative stress one of the proposed mechanisms, the objective is to determine the effect of supplementation with β-carotene to type 2 diabetics and healthy individuals, on iron metabolism, oxidative balance, and antioxidant plasma capacity, using doses similar to the daily nutritional requirement.

DETAILED DESCRIPTION:
Type 2 diabetes is a chronic, multifactorial disease, and oxidative stress one of the pathophysiological mechanisms associated with its appearance and development. The objective was to determine the effect of supplementation with β-carotene to type 2 diabetics and healthy individuals, on iron metabolism, oxidative balance, and antioxidant plasma capacity, using doses similar to the daily nutritional requirement.

A total of 117 volunteers participated in the study. Type 2 diabetics (34) and healthy individuals (24), received 6 mg β-carotene for 45 d, and were compared to similar non-supplemented diabetic (33) and control (26) groups. Blood samples were taken at the beginning, end and 30 days after finishing supplementation, to determine hemoglobin, hematocrit unsaturated iron binding capacity, total iron binding capacity, transferrin saturation, ferritin, glycemia, glycosylated hemoglobin, cholesterol, triglycerides, HDL, LDL, oxidized LDL, copper, zinc, TBARS, FRAP, nitrites, GPx, SOD, folates, retinol and β-carotene.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnose of Type 2 diabetes mellitus of at least 5 years of diagnosis, in treatment with oral hypoglycemics Patients in regular control (once a month) in the Hospital

Exclusion Criteria:

* Hospitalized patient
* Diabetic patient with diabetes related acute complications (ketoacidosis, hyperosmolar coma)in the 3 months previous to the study.
* Individuals with infections that required antibiotics in the 3 weeks previous to the study.
* Individuals with antibodies anti-insulin, autoimmune diseases or in treatment with immunosuppressive drugs.
* Individuals with viral infections such as hepatitis B, hematological, renal or hepatic diseases.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in oxidative status | Time 0, 45 days and 75 days after supplementation

SECONDARY OUTCOMES:
Hemoglobin and hematocrit | Time 0, 45 days and 75 days after supplementation
Ferritin | Time 0, 45 days and 75 days after supplementation
  Enzyme linked immunosorbent assay (ELISA) with monoclonal antibodies
Iron metabolism markers | Time 0, 45 days and 75 days after supplementation
  Serum iron, total iron binding capacity (TIBC) and unsaturated iron binding capacity (UIBC) were determined by the methods proposed by the International Committee of Standardization of Hematology.
Blood Chemistry | Time 0, 45 days and 75 days after supplementation
  Glycemia, triglycerides, total cholesterol, LDL, and HDL were determined automatically in a Ciba Corning 550 Express autoanalizer, using classic enzymatic methods for the determination of these variables.
Glycosylated Hemoglobin | Time 0, 45 days and 75 days after supplementation
  It was determined using a commercial kit (Bioscience, Caracas, Venezuela),
Oxidized LDL | Time 0, 45 days and 75 days after supplementation
  Analyzed by a solid phase two-site enzyme immunoassay from Mercodia (Sweden), which contains 2 monoclonal antibodies directed against separated antigenic determinants on the oxidized apolipoprotein B molecule.
Thiobarbituric Acid Reactive substances (TBARS) | Time 0, 45 days and 75 days after supplementation
  Were detected by the quantification of malondialdehyde present in the sample, by reacting 2 molecules of thiobarbituric acid with 1 molecule of malondialdehyde, which produces an abduct that is detected at 535 mn.
Ferric Reducing ability of Plasma (FRAP). | Time 0, 45 days and 75 days after supplementation
  Measured after 4 and 10 min incubation, was used to determine the ability of plasma to reduce iron from ferric to ferrous state, based on the formation of a triazine-Fe+3 complex, that when reduced to Fe+2, generate a change in color that is measured at 593 nm.
Activities of the enzymes superoxide dismutase (SOD) and glutathione peroxidase (GPx). | Time 0, 45 days and 75 days after supplementation
  Determined by commercial kits (Cayman Chemicals, Pittsburg) following the recommended protocols
Serum zinc and copper. | Time 0, 45 days and 75 days after supplementation
  By flame atomic absorption spectrophotometry
β-carotene. | Time 0, 45 days and 75 days after supplementation
  It was determined by HPLC, with a reverse fase C18 column.
Serum retinol | Time 0, 45 days and 75 days after supplementation
  It was determined by HPLC, with a reverse fase C18 column, as an indirect measure of betacarotene metabolism.
Serum nitrites | Time 0, 45 days and 75 days after supplementation
  Were determined as an indirect measure of the concentration of nitric oxide, since nitrites are the stable end products of its degradation. Nitrates were reduced to nitrites by activated cadmium. Then sulfanilamide and nitrites generate a chromophore that reacts with naftilethylenediamine, to generate a product visible at 540 nm.
Serum and erythrocyte folates. | Time 0, 45 days and 75 days after supplementation
  The method is based in the folate-dependent controlled growth of a Lactobacillus strain that is measured spectrophotometrically and quantified against a standard curve.

CONTACTS AND LOCATIONS:
Overall Officials: Maria N Garcia-Casal, PhD, Study Director — Instituto Venezolano de Investigaciones Cientificas; Jose M Moreno, PhD, Principal Investigator — Instituto Venezolanode Investigaciones cientificas
Locations (1):
- Hospital Baudilio Lara, Barquisimeto, Lara, Venezuela

REFERENCES:
- [Background] Ford ES, Cogswell ME. Diabetes and serum ferritin concentration among U.S. adults. Diabetes Care. 1999 Dec;22(12):1978-83. doi: 10.2337/diacare.22.12.1978. PMID 10587829
- [Background] Ford ES, Mokdad AH, Giles WH, Brown DW. The metabolic syndrome and antioxidant concentrations: findings from the Third National Health and Nutrition Examination Survey. Diabetes. 2003 Sep;52(9):2346-52. doi: 10.2337/diabetes.52.9.2346. PMID 12941775
- [Background] Sugiura M, Nakamura M, Ikoma Y, Yano M, Ogawa K, Matsumoto H, Kato M, Ohshima M, Nagao A. The homeostasis model assessment-insulin resistance index is inversely associated with serum carotenoids in non-diabetic subjects. J Epidemiol. 2006 Mar;16(2):71-8. doi: 10.2188/jea.16.71. PMID 16537987
- [Background] Song Y, Cook NR, Albert CM, Van Denburgh M, Manson JE. Effects of vitamins C and E and beta-carotene on the risk of type 2 diabetes in women at high risk of cardiovascular disease: a randomized controlled trial. Am J Clin Nutr. 2009 Aug;90(2):429-37. doi: 10.3945/ajcn.2009.27491. Epub 2009 Jun 2. PMID 19491386
- See also: American Diabetes Association — http://www.diabetes.org